CLINICAL TRIAL: NCT01293331
Title: Prospective Surveillance of Febrile Illness for Dengue-Endemic Areas in Latin America
Brief Title: Study of Febrile Illness for Dengue-Endemic Areas in Latin America
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: CYD35; U1111-1112-8481 (Other: WHO)
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Dengue Fever; Fever
Keywords: Dengue Fever Fever Seroprevalence
MeSH Terms: conditions — Dengue; Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Cohort (Case ): Participants will be examined for fever in dengue endemic regions

SUMMARY:
The purpose of this study is to detect acute febrile episodes and dengue infection in five Latin American countries to assess dengue seroprevalence.

Primary objectives:

* To identify acute febrile episodes among the cohort in order to detect the presence of dengue infection.
* To describe the dengue seroprevalence among the cohort at baseline and at the end of the study.

DETAILED DESCRIPTION:
All participants will make two visits to a study site, an enrollment visit and a termination visit. Additional visits will be made if febrile episodes occur: an acute visit and a convalescent visit. Participants or their parents/guardians will be contacted weekly to monitor the occurrence of febrile episodes and ensure appropriate assessment and care.

No vaccine will be provided or administered in this study

ELIGIBILITY:
Inclusion Criteria :

* Aged 9 to 16 years on the day of inclusion and resident of the site zone
* Participant in good health, based on medical history and physical examination
* Assent form has been signed and dated by the participant (if required by local regulations), and informed consent form has been signed and dated by the parent(s) or another legally acceptable representative (and by the participant and/or an independent witness if required by local regulations)
* Participant able to attend all scheduled visits and to comply with all study procedures

Exclusion Criteria :

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding enrollment
* Planned participation in another clinical trial during the present study period
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroids therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported seropositivity for Human Immunodeficiency Virus (HIV) infection
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion
* Current alcohol abuse or drug addiction that may interfere with the participant's ability to comply with study procedures
* Receipt of blood or blood-derived products in the past 3 months
* Receipt of any vaccine in the 4 weeks preceding the day of enrollment except for pandemic influenza vaccination, which may be received at least 2 weeks before enrollment
* Planned receipt of any vaccine in the 4 weeks following enrollment
* Deprived of freedom by administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Identified as employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members (i.e., immediate, husband, wife and their children, adopted or natural) of the employees or the Investigator.

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants aged 9 to 16 years in 4 countries in Latin America: Brazil, Mexico, Colombia and Puerto Rico
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Identification of acute febrile episodes in the cohort | Up to 18 months after study entry
Detection of confirmed or probable dengue infection in the cohort | Up to 18 months after study entry

CONTACTS AND LOCATIONS:
Overall Officials: Regional Director, Study Director — Sanofi Pasteur SA.
Locations (18):
- Brazil (4):
  - Campo Grande
  - Goiânia
  - Natal-RN
  - Vitória
- Colombia (8):
  - Acacias Meta
  - Aguazul (Casanare)
  - Bogotá
  - Calarco (Quindio)
  - Girardot (Cundinamarca)
  - La Tebaida (Quindio)
  - Montenegro (Quindio)
  - Yopal (Casanare)
- Mexico (4):
  - Minatitlán, Veracruz Mexico
  - Veracruz, Veracruz Mexico
  - Municipio de Cd. Mante Tamaulipas
  - Quintana Roo
- Puerto Rico (2):
  - Guayama, Puerto Rico
  - San Juan, Puerto Rico

REFERENCES:
- [Result] Dayan G, Arredondo JL, Carrasquilla G, Deseda CC, Dietze R, Luz K, Costa MSN, Cunha RV, Rey LC, Morales J, Reynales H, Miranda M, Zambrano B, Rivas E, Garbes P, Noriega F. Prospective cohort study with active surveillance for fever in four dengue endemic countries in Latin America. Am J Trop Med Hyg. 2015 Jul;93(1):18-23. doi: 10.4269/ajtmh.13-0663. Epub 2015 May 26. PMID 26013373
- See also: Related Info — http://www.sanofipasteur.com